CLINICAL TRIAL: NCT04051866
Title: Effectiveness of Non-surgical Periodontal Treatment on HbA1c Levels in a Patient With Type 2 Diabetes Mellitus in Primary Care: Randomized Clinical Trial
Brief Title: Effectiveness of Non-surgical Periodontal Treatment on HbA1c Levels in a Patient With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a Cochrane review whose authors conclude that further trials evaluating periodontal treatment versus no treatment/usual care are unlikely to change the overall conclusion reached in this review.
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Juan Ignacio Ropero Pires, Dentist. Principal investigator, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI 20/18
Record Dates: First submitted 2019-07-16; First posted 2019-08-09 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Chronic Periodontitis; Diabetes Mellitus, Type 2
Keywords: Dentist; Primary Health Care; Chronic Periodontitis; Diabetes Mellitus, Type 2; Root planing; Dental Scaling
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2 | interventions — Root Planing

STUDY DESIGN:
Intervention Model Description: The sample size has been calculated to estimate a difference of at least 0.4% units between groups in the change of HbA1c at 12 months.
  By means of a list of the patients assigned in the usual practice to each participating dentist, who meets the inclusion criteria, and they will be contacted in the resulting order after carrying out a randomization of each list.
  Once it has been confirmed that it meets the inclusion criteria and accepted the participation in it, a simple random assignment, with balanced groups, will be used, automatically implemented in the electronic data collection notebook.
  The intervention can not be masked, however the main result is measured through an analytical parameter (HbA1c), minimizing the possibility of information bias.
  To reduce the possible variability due to the different observers, a training and calibration session will be developed.
Masking Description: Intervention can't be masked. Statistician conducting the analysis will not know to which study arm a given patient has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Usual care (provided in Primary Health Care Centres) Oral hygiene instructions
  Interventions: Other: Oral hygiene instructions
- Intervention (Experimental): Usual care (provided in Primary Health Care Centres) Non-surgical periodontal treatment: Scaling and root planing (SRP) Oral hygiene instructions
  Interventions: Procedure: Non-surgical periodontal treatment: Scaling and root planing (SRP); Other: Oral hygiene instructions

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment: Scaling and root planing (SRP) — Removal of dental plaque and dental calculus from the surface of a tooth, from the surface of a tooth apical to the gingival margin accumulated in periodontal pockets, or from the surface coronal to the gingival margin.
  Arms: Intervention
Other: Oral hygiene instructions — Education for individual health regarding peridontal disease and its association with diabetes, as well as oral hygiene instructions that include the modified Bass technique, use of interproximal brushes and dental floss

SUMMARY:
This study evaluates the effectiveness of an intervention, non-surgical periodontal treatment (SPR), in patients with poorly controlled type 2 diabetes mellitus and moderate-severe periodontal disease aimed at reducing HbA1c levels at 12 months compared with the usual practice in Primary Health Care.

DETAILED DESCRIPTION:
Design: Pragmatic cluster randomized clinical trial with 12 months follow-up. Unit of randomization: dentist. Setting: Primary Health Care Centers in one Spanish region (Madrid) Population: Patients ≥ 35 years of age with moderate-severe periodontal disease and diagnosed with type 2 diabetes with por control (HbA1c > 7,5). N=288 patients (144 in each arm) will be recruited by dentist before randomization.

Intervention: Both groups will receive education on oral hygiene measures. The experimental group will receive the non-surgical periodontal treatment at the beginning of the study and the control group at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes (code CIAP-2 T90)
* With at least one determination of HbA1c in the last 3 months HbA1c> 7.5%
* No changes in hypoglycemic or insulin treatment in the last 3 months.
* With generalized moderate-severe chronic periodontal disease.
* Presence of at least 16 natural teeth.
* Informed consent.

Exclusion Criteria:

* Patients with basic systemic diseases with oral involvement (autoimmune diseases of oral involvement: oral lichen planus, lupus, pemphigus, pemphigoid)
* Limited life expectancy.
* Urgent diabetic complications in the 30 days prior to the study.
* They need extensive oral treatment: fistulous trajectories, cellulitis, pulpitis or other oral infections.
* Pregnant, with desire for pregnancy in the 12 months of study or breastfeeding.
* That they have received periodontal treatment in the last 6 months.
* That they have received antibiotic and / or anti-inflammatory regimen continued at least in the last 4 weeks prior to the study (except low doses of acetylsalicylic acid).
* In treatment with corticosteroids or immunosuppressive drugs.
* On dialysis or risk of bleeding (anticoagulant treatment).
* Dependent on alcohol.
* Patients who require antibiotic prophylaxis for the realization of SPR.
* Patients with uncontrolled systemic diseases (with the exception of diabetes): cardiovascular, lung, liver, kidney disease in advanced stages or neoplasms.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-02 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin A (HbA1c) | Change from baseline HbA1c score at 6 and 12 months
  Products of non-enzymatic reactions between GLUCOSE and HEMOGLOBIN A, occurring as a minor fraction of the hemoglobin components of human erythrocytes. Glycated hemoglobin A is used as an index of the average blood sugar level over a lifetime of erythrocytes.
  Glycated hemoglobin (A1C) goals in patients with diabetes should be tailored to the individual, balancing the demonstrated benefits with regard to prevention and delay in microvascular complications with the risk of hypoglycemia. A reasonable goal of therapy might be an A1C value of ≤7.0 percent for most medication-treated patients (using an assay aligned to the Diabetes Control and Complications Trial in which the upper limit of normal is 6.0 percent). Glycemic targets are generally set somewhat higher (eg, <8 percent) for older adult patients and those with comorbidities or a limited life expectancy and little likelihood of benefit from intensive therapy.

SECONDARY OUTCOMES:
Probing depth | basal measurement, at 6 and 12 months
  The measured distance from the free end of the gingival margin to the bottom of the periodontal pocket. Measurement in milimetres. Depths greater than 3 mm can be associated with "attachment loss" of the tooth to the surrounding alveolar bone, which is a characteristic found in periodontitis.
Glomerular filtration | basal measurement, at 6 and 12 months
  The volume of water filtered out of plasma through glomerular capillary walls into Bowman's capsules per unit of time
Quality of life of patients: EuroQol 5D-5L questionnaire | Basal measurement, at 6 and 12 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. Each of the 5 dimensions comprising the EQ-5D descriptive system is divided into 5 levels of perceived problems: 1: no problem. 2: slight problems 3: moderate problems. 4: severe problems. 5: extreme problems
Physical activity (IPAQ questionnaire) | Basal measurement, at 6 and 12 months
  IPAQ was developed for comparable and valid measures of physical activity within and between countries, across various life domains. Three levels are proposed: Category 1: Low: This is the lowest level of physical activity. Those individuals who not meet criteria for categories 2 or 3 are considered low/inactive. Category 2: Moderate: Any one of the following 3 criteria:
  * 3 or more days of vigorous activity of at least 20 minutes per day
  * 5 or more days of moderate-intensity activity or walking of at least 30 minutes per day
  * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-min/week.
  Category 3: High: Any one of the following 2 criteria:
  * Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week
  * 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET-minutes/week
Diet questionnaire (MEDAS) | Basal measurement, at 6 and 12 months
  The MEDAS is a 14-item questionnaire that asks participants to report the usual frequency of consumption or the amount consumed of 12 main components of MedDiet and two eating habits related to MedDiet. Each of the 14 items is scored 1 or 0, depending on whether the participants adhere to each MedDiet component or not. If these conditions were not met, an item was assigned a score of 0. The resulting MedDiet score of MEDAS varied from 0 to 14. Photographs of portions and portion sizes were used, as appropriate, to facilitate completion of MEDAS TOTAL SCORE: < 9 low adhesion; > = 9 good adhesion
Therapeutic adherence questionnaire (Morisky-Green) | Basal measurement, at 6 and 12 months
  It consists of a series of four contrast questions with dichotomous answer (yes / no), which reflects the patient's behavior regarding compliance. It is intended to assess whether the patient adopts correct attitudes regarding the treatment for his illness; It is assumed that if the attitudes are incorrect, the patient is non-compliant. It has the advantage of providing information on the causes of the breach. The patient is considered as compliant if he answers the four questions correctly.
Cost-utility | At 12 months
  The calculation of benefits will be made in the form of QALYs accounting for the total profit in profits, measured with the EuroQol 5D-5L in the intervention group
Gingival Recession | basal measurement, at 6 and 12 months
  Exposure of the root surface when the edge of the gum (GINGIVA) moves apically away from the crown of the tooth. Measurement in milimetres. Greater gingival recession can be associated with "attachment loss" of the tooth to the surrounding alveolar bone, which is a characteristic found in periodontitis.
Clinical attachment level | basal measurement, at 6 and 12 months
  The distance from the cementoenamel junction to the bottom of the periodontal pocket. Measurement in millimetres. Greater clinical attachment level can be associated with "attachment loss" of the tooth to the surrounding alveolar bone, which is a characteristic found in periodontitis.
Gingival Probing bleeding | basal measurement, at 6 and 12 months
  Measured as the percentage of sites with blood present at the probing (present: if it occurred within 30 seconds of the probing. Absent: if no bleeding occurred). Greater gingival probing bleeding can be associated with "Inflammation of gum tissue", which is a characteristic found in periodontitis.

CONTACTS AND LOCATIONS:
Overall Officials: María Trinidad García Vázquez, Dentist, PhD, Principal Investigator — Gerencia de Atención Primaria
Locations (1):
- Gerencia de Atención Primaria, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No